CLINICAL TRIAL: NCT06529549
Title: A Prospective, Open-label, Single-arm Study on the Efficacy and Safety of Organoid-Based Drug Sensitivity Screening to Guide the Treatment of mCRPC Patients With Bone Metastasis Progressed After First-line Treatment
Brief Title: Efficacy and Safety of Organoid-Based Drug Sensitivity Screening to Guide the Treatment of mCRPC Patients Progressed After First-line Treatment
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Professor, Sun Yat-sen University
Other Study IDs: 2024-FXY-231
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Organoid-Based Drug Sensitivity Screening: Organoid culture and drug sensitivity screening
  Interventions: Other: Organoid-Based Drug Sensitivity Screening

INTERVENTIONS:
Other: Organoid-Based Drug Sensitivity Screening — Residual tissue of bone metastatic sites from biopsies for genetic testing will be collected to culture organoid and perform drug sensitivity screening

SUMMARY:
This observational study aims to learn about the effects and safety of organoid-based drug sensitivity screening in mCRPC patients with bone metastases that progressed after first-line treatment. The main question it seeks to answer is:

Do doctors choose treatment agents based on organoid-based drug sensitivity screening results for mCRPC patients, resulting in a better response?

Participants already took bone metastasis biopsies for genetic testing based on current clinical guidelines. This study only takes residual tissue from biopsies for organoid culture.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Adult males from 18 to 75 years age.
3. History of histologically or cytologically confirmed adenocarcinoma
4. Documented evidence of metastatic castration resistant prostate cancer (mCRPC) and progressed after first-line treatment at mCRPC.
5. Evidence of target lesion in imaging studies.
6. ECOG performance status 0-1
7. Estimated survival≥12 weeks

Exclusion Criteria:

1. Do not meet the inclusion criteria.
2. Under any other anti-tumor therapy like chemotherapy and/or immunotherapy.
3. Receiving organ transplantation in the last 3 months.
4. Participants with autoimmune diseases or history of HBV, HCV or HIV infection (acute).
5. Participants with pneumonia.
6. Severe concurrent illness or co-morbid disease that would make the subject unsuitable for enrolment
7. Unwilling and unable to provide informed consent.
8. Patients who are judged unsuitable for clinical trial participation by the investigators.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mCRPC patients with bone metastases and progressed after first-line treatment of mCRPC stage
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2027-07-23 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) Response Rate | From enrollment to primary completion of study (up to approximately 3 years)
  Proportion of patients with a 50% decrease in PSA from baseline

SECONDARY OUTCOMES:
Radiologic Progression-free Survival (rPFS) | 3 years
  Radiologic progression-free survival will be assessed from the time of the first dose to radiologic disease progression or death from any cause, whichever comes first.
Objective Response Rate (ORR) | From enrollment to primary completion of study (up to approximately 3 years)
  Proportion of patients in complete remission (CR) plus partial remission (PR)
Duration of Response (DOR) | From enrollment to primary completion of study (up to approximately 3 years)
  Time from the start of the first assessment of the tumor as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
Overall Survival (OS) | From enrollment to primary completion of study (up to approximately 3 years)
  Time between the start of treatment and death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided